CLINICAL TRIAL: NCT01840007
Title: Pilot Study Evaluating the Efficacy and Safety of Metformin in Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-PP-17; 2010-024322-38 (EudraCT Number)
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2022-11-29 (Actual); Status verified 2013-02

CONDITIONS: Metastatic Melanoma (Stage IIIC Non-résécable or no Surgically Curable or Stage IV With Classification AJCC)
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Metformin (Experimental): The chosen posology is 2540 mg/day of metformin-base so 3 tablets/day of Glucophage ® 1000.
  Patients should take 3 tablets/day at the rate of 1tablet in morning, noon and evening to favor the absorbtion and reduce the risk of gastrointestinal intolerance. In case of missed dose, patients will be allowed to take 2 tablets on the next grip. The drug will be presented in its officinale form of Glucophage ® 1000 with specifications indicated in the Vidal dictionary. It will be provided each month, to patient, 3 boxes of 30 tablets of Glucophage ® 1000. The patient will be asked to rate each day, on a calendar, the number of tablets of Glucophage ® 1000 effectively taken. It will also ask to the patient to bring back used boxes of Glucophage ® 1000 to count any tablets not taken.
  Interventions: Drug: Metformin Group

INTERVENTIONS:
Drug: Metformin Group — The chosen posology is 2540 mg/day of metformin-base so 3 tablets/day of Glucophage ® 1000.
  Patients should take 3 tablets/day at the rate of 1tablet in morning, noon and evening to favor the absorbtion and reduce the risk of gastrointestinal intolerance. In case of missed dose, patients will be allowed to take 2 tablets on the next grip. The drug will be presented in its officinale form of Glucophage ® 1000 with specifications indicated in the Vidal dictionary. It will be provided each month, to patient, 3 boxes of 30 tablets of Glucophage ® 1000. The patient will be asked to rate each day, on a calendar, the number of tablets of Glucophage ® 1000 effectively taken. It will also ask to the patient to bring back used boxes of Glucophage ® 1000 to count any tablets not taken.

SUMMARY:
In western countries, melanoma represents a major mistake of public health by its frequency, lethality and the increasing of incidence. Surgery can cure melanoma diagnosed very early. In other cases, it exists a risk of recurrence of lymph node and visceral. At the stage of visceral metastases, the prognosis of melanoma is catastrophic, with a median survival of 6 months. Indeed, the reference chemotherapy by dacarbazine induces a very limited response rate of 10-20%, the ipilimumab which has been authorized in the second intention, has a response rate of 10%, and other available treatments don't have a superior efficiency. Metformin is an oral antidiabetic of biguanides family which acts by inducing the activation of AMPK, a molecule which is inactivated in many cancers including the melanoma. In agreement with these data, several preclinical studies suggested that metformin has antineoplastic activity. In the case of melanoma, a study published recently has showed that metformin inhibits proliferation of melanoma cells in vitro and we confirmed for our part these results in our laboratory (INSERM U895).

ELIGIBILITY:
Inclusion Criteria:

* Major patients with metastatic melanoma (stage IIIC non-résécable or no surgically curable or stage IV with classification AJCC) in progression after a first-line of treatment by vemurafenib or chemotherapy, and non-eligible or non-responders to ipilimumab.

Metastases measurable by RECIST criteria. Hematologic, renal and hepatic appropriate functions. Negative pregnancy test.

Exclusion Criteria:

* Patients with symptomatic brain metastases and Performans Status (PS)>2. Patients with carcinomatous meningitis. Pregnant or breathfeeding women. Patients with a contraindication to the metformine. HIV infection, active infection with HBV or HCV. Patients already treated with metformin in the context of diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08-30 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2015-11-18 (Actual)

PRIMARY OUTCOMES:
Response rate | Once time after 6 months of treatment by metformine
  The primary evaluation criteria is the response rate (response rate, RR) defined by the ratio between the total number of patients with a complete response (complete response, CR) or partial (partial response, PR) and the total number of patients in the study. Partial or complete responses will be defined by RECIST 1.1 (15) criteria :
  * Complete response: disappearance of all targets lesions
  * Partial response: decrease of at least 30% of the sum of the biggest diameters of each target lesion All others patients, including those for who the response couldn't be measured, will be considered non-responders.

SECONDARY OUTCOMES:
the overall survival, the survival without progress (PFS), the tolerance, and the quality of life. | 6 times
  * Overall survival (OS) is defined by the duration (number of days) between the start of treatment (J1) and the date of death from anything.
  * Progression-free survival (PFS) is defined by the duration (number of days) between the start of treatment (J1) and the observation of a progression or death. Tumor progression is defined by an increase of at least 20% of the sum of the biggest diameters of each target lesion.
  * The duration of the response is determined by the time (in days) between the date (visit) which is recorded a response to the treatment (complete or partial) and the date (visit) which is recorded an increase or the date of death.
  * To evaluate the quality of life, a questionnaire EORTC QLQ-C30 version 3 (16), validated in French, will be completed by the patient at visits V1 (J1), V3 (M2), V5 (M4) and V7 (M6) (Annex X).

CONTACTS AND LOCATIONS:
Overall Officials: BAHADORAN Philippe, PHD, Principal Investigator — Service de Dermatologie - Hôpital de l'Archet - CHU de Nice
Locations (2):
- France (2):
  - Bahadoran, Nice, Alpes-Maritimes
  - MORTIER Laurent, Lille, Nord